CLINICAL TRIAL: NCT02341950
Title: Evaluating the Effectiveness of a Serious Game to Enhance Self-Management Skills Among Adolescents and Young Adults With Spinal Cord Dysfunction
Brief Title: Clinical Trial of a Serious Game for Individuals With SCI/D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Meade, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UM-RERC-82972
Record Dates: First submitted 2014-12-16; First posted 2015-01-19 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Spinal Cord Injury; Spinal Cord Involvement; Spina Bifida; Transverse Myelitis; Polio and Post-polio Syndrome; Syringomyelia; Spinal Stenosis; Spinal Neoplasms; Spinal Cord Diseases
Keywords: videogame; health; behavior; mobile; spinal; cord; dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Dysraphism; Myelitis, Transverse; Postpoliomyelitis Syndrome; Syringomyelia; Spinal Stenosis; Spinal Neoplasms; Spinal Cord Diseases; Behavior; Cone-Rod Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCI Hard (Experimental): This arm plays the SCI HARD game
  Interventions: Behavioral: SCI Hard
- Control (No Intervention): Plays an alternate, publicly available game

INTERVENTIONS:
Behavioral: SCI Hard — The game SCI Hard is designed to enhance self-management skills in individuals with spinal cord injury
  Arms: SCI Hard

SUMMARY:
This study will evaluate the efficacy of a newly developed serious game, SCI HARD, to enhance self-management skills, self-reported health behaviors, and quality of life among adolescents and young adults with spinal cord injury and disease (SCI/D). SCI HARD was designed by the project PI, Dr. Meade, in collaboration with the UM3D (University of Michigan three dimensional) Lab between 2010 and 2013 with funding from a NIDRR (National Institute on Disability and Rehabilitation Research) Field Initiated Development Grant to assist persons with SCI develop and apply the necessary skills to keep their bodies healthy while managing the many aspects of SCI care. The study makes a unique contribution to rehabilitation by emphasizing the concepts of personal responsibility and control over one's health and life as a whole. By selecting an innovative approach for program implementation, we also attempt to address the high cost of care delivery and lack of health care access to underserved populations with SCI/D living across the United States (US).

H1: SCI Hard participants will show greater improvements in problem solving skills, healthy attitudes about disability, and SCI Self-efficacy than will control group members; these improvements will be sustained over time within and between groups.

H2: SCI Hard participants will endorse more positive health behaviors than control group members; these improvements will be sustained over time within and between groups.

H3: SCI Hard participants will have higher levels of QOL than control group members; these differences will be sustained over time within and between groups.

H4: Among SCI Hard participants, dosage of game play will be related to degree of change in self-management skills, health behaviors and QOL.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of a newly developed serious game, SCI HARD, to enhance self-management skills, self-reported health behaviors, and QOL among adolescents and young adults with spinal cord injury and disease (SCI/D). SCI HARD was designed by the project PI, Dr. Meade, in collaboration with the UM3D Lab between 2010 and 2013 with funding from a NIDRR (National Institute on Disability and Rehabilitation Research) Field Initiated Development Grant to assist persons with SCI develop and apply the necessary skills to keep their bodies healthy while managing the many aspects of SCI care. The study makes a unique contribution to rehabilitation by emphasizing the concepts of personal responsibility and control over one's health and life as a whole. By selecting an innovative approach for program implementation, we also attempt to address the high cost of care delivery and lack of health care access to underserved populations with SCI/D living across the United States (US).

BACKGROUND AND LITERATURE REVIEW As defined by the computer gaming industry, a serious game is "a game designed for a primary purpose other than pure entertainment." Serious games based on development of self-management skills have been developed for asthma, diabetes, safe sex negotiation, and promoting nutrition and physical activities. They have been effective in improving self-care, increasing self-efficacy, reducing symptoms, minimizing secondary conditions, reducing emergency room visits and decreasing health care costs.

The game application being assessed in this project is based on the self-management principles and specifically on the Health Mechanics Program, an evidence-based self-management program which was developed by Dr. Meade. Many of the individuals who sustain traumatic SCI are from the millennial generation. While the mean age for individuals with SCI is 40.2 years old, approximately half are in the 16 to 29 age range at the time of injury. Younger patients with traumatic SCI are overwhelmingly male, many of whom need medical care for the first time in their lives. These individuals are likely to be single (never-married) and many have a high-school education or less. A significant component of this group was injured through participation in high-risk behaviors or acts of violence; the group tends to have lower literacy levels and fewer resources, with many being from ethnic and racial minority backgrounds.

As previously discussed, individuals in this group, tend to have a high degree of technical sophistication which can be leveraged to promote the transfer of knowledge and self-management skills. In particular, games that can be downloaded and played on a mobile platform, such as a smartphone, are likely to be accessed and played by members of this group.

Data from the Pew Internet and American Life Project indicates that most Americans age 16 to 24 play computer or electronic games - including 97% of American teenagers and 81% of adults 18 to 29 years old. African Americans appear equally likely to play electronic games as Non-Hispanic Whites (both 51%) while English-Speaking Hispanics appear more likely to do so (63%; though that was attributed to the youth of the group). While most adult gamers play on the computers (73%), teens and young adults are increasingly playing on portable gaming devices (62%) and cell phones (50%). African Americans and Hispanics are more likely than non-Hispanic, Whites to play games on smaller, mobile gadgets. 55% of teens own a portable gaming device, 74% own an iPod or MP3 player, and 60% have a desktop or laptop computer.

Data from a recent survey conducted by Dr. Meade and her colleague confirms the use of technology by individuals with SCI. They sent a mail survey to the population of individuals with SCI ages 8 and older who were identified as being treated at the U-M within the past 10 years. Among those individuals who appeared to have valid addresses (n=780), approximately 40% (n=317) responded. While most of these individuals owned a computer and many owned other types of devices, more than half of 13 to 29 year olds owned or used a mobile device that could be used for gaming (e.g., iPad, iPhone, Android table / phone).

INTERVENTION SCI HARD was designed based on the needs and strengths of individuals with SCI/D while being responsive to identified gaps and challenges in health care provision in this population. Current theories of health behavior and standard practices for game development shaped its development. In particular, we referred to the previously described model proposed by Ritterband et al. for behavior change using internet interventions and prioritized fun and engagement in the design process. The program focuses on enhancing skills, encouraging positive health behaviors and empowering people within their own environments, recognizing that people have different resources and abilities. By teaching skills to better manage health, this self-management program should not only reduce the occurrence of complications but should also promote higher levels of social integration and QOL. In particular, playing the game should allow players to recognize the consequences of their behaviors as actions and inactions are tied to visible results and substantial changes in statistics.

As currently developed, SCI Hard is available on both IOS (Apple Mobile Operating System) and Android platforms. Play time is approximately 5 hours and requires individuals to be able to successfully manage their health before they will be able to complete all levels.

Purpose and Objectives The overall purpose is to evaluate the effects of the serious game SCI Hard on self-management skills, positive health behaviors and QOL. The program specifically targets adolescents and young adult with SCI/D.

Objectives are: 1) to improve self-management skills, including problem-solving, attitude about disability, and self-efficacy for managing health; 2) to increase performance of recommended health management behaviors; 3) to improve QOL; and 4) to determine the extent that dosage of game play impacts changes in any of these factors. .

All hypotheses posit that, following the intervention, differences will exist such that participants in the SCI Hard will show more positive outcomes than the control group members (an assessment of between group differences) and that these differences will be sustained over time (an assessment of within and between group differences). It is expected that, for the intervention group, degree of engagement with the game (or dosage or play time) will influence degree of improvements, thus our interest in examining within group differences.

Research Hypotheses H1: SCI Hard participants will show greater improvements in problem solving skills, healthy attitudes about disability, and SCI Self-efficacy than will control group members; these improvements will be sustained over time within and between groups.

H2: SCI Hard participants will endorse more positive health behaviors than control group members; these improvements will be sustained over time within and between groups.

H3: SCI Hard participants will have higher levels of QOL than control group members; these differences will be sustained over time within and between groups.

H4: Among SCI Hard participants, dosage of game play will be related to degree of change in self-management skills, health behaviors and QOL.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 13 and 29
* have a spinal cord dysfunction
* have access to a mobile device on which they can download and play the game
* be English-speaking.

Exclusion Criteria:

* high degrees of emotional distress, suicidal intent, or anxiety (as determined by the Patient Health Questionnaire-Depression Module (PHQ-9) and Generalized Anxiety Disorder-7(GAD-7)). Individuals will also be required to answer questions to confirm that they understand the study as part of the informed consent process.

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Appraisals of Disability: Primary and Secondary Scale (ADAPSS) (used to assess change over time) | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in six dimensions of appraisal: fearful despondency, overwhelming disbelief, determined resolve, growth and resilience, negative perceptions of disability, and personal agency.
Change in scores on the Disability Management Self-Efficacy Scale - Short | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in the extent that the person with a SCI feels they can manage their health and keeping it from interfering with their life
Change in scores on the Effective Consumer Scale | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in how effective people are at dealing with their chronic condition and making decisions about their health care".

SECONDARY OUTCOMES:
Frequency & Interval of game play | Information about dosage of play
  Transmitted wirelessly while participant is playing the game
Change in scores on the SCI/D Self-monitoring inventory | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in self-monitoring
Change in scores on the Social Problem Solving Inventory - Revised: Short Form | change in scores on the SPSI-R from baseline (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in 4 dimensions of problem solving: negative
Change in scores on the Craig Handicap Assessment and Reporting Technique - Short Form (CHART-SF) | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in impairments and disabilities that result in handicaps in the years after initial rehabilitation.
Change in scores on the WHOQOL-BREF (World Health Organization Quality of Life) | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in specific domains of health related Quality of Life
Change in scores on the Spinal Cord Injury Lifestyle Scale | change scores at 1 months and 3 months (baseline to 1 month; baseline to 3 months; 1 month to 3 months)
  Used to assess change over time in health behaviors that may have an indirect effect on complications

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Meade, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data is not planned to be released.